CLINICAL TRIAL: NCT04198519
Title: Effects of Weight Loss on Vascular Function in Obese Individuals With Poor Cardiovascular Health
Brief Title: Effects of Weight Loss on Vascular Function in Obese Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mario Fritsch Neves (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor-Investigator, Mario Fritsch Neves, Clinical Professor, Hospital Universitario Pedro Ernesto
Organization: Hospital Universitario Pedro Ernesto (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WL-50
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Cardiovascular diseases; Sleep Apnea Syndromes; Arterial stiffness; Endothelial dysfunction
MeSH Terms: conditions — Obesity; Weight Loss; Cardiovascular Diseases; Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Prospective
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants do not know if they are classified as poor or intermediate/ideal cardiovascular health.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Poor Cardiovascular Health (Active Comparator): Cardiovascular health is said to be ideal by the presence of optimal health behaviors (non-smokers, adequate BMI, physical activity level and healthy eating pattern) and ideal health factors (blood pressure, total cholesterol and blood glucose). Poor cardiovascular health is considered for two or less metrics.
  Interventions: Other: Weight Loss
- Ideal-intermediate Cardiovascular Health (Active Comparator): Cardiovascular health is said to be ideal by the presence of optimal health behaviors (non-smokers, adequate BMI, physical activity level and healthy eating pattern) and ideal health factors (blood pressure, total cholesterol and blood glucose). Ideal cardiovascular health is considered for those with five or more metrics within this qualification, and intermediate for the presence of three or four metrics.
  Interventions: Other: Weight Loss

INTERVENTIONS:
Other: Weight Loss — The total energy value (TEV) of the diet prescribed for each study participant will be determined by subtracting 800 kcal / day from the total daily energy expenditure, which will be based on Dietary Reference Intake (DRI) recommendations. The distribution of macronutrients will be as follows: protein 15 to 20% of TEV, lipids 25 to 30% of TEV and carbohydrates 50 to 60% of TEV.

SUMMARY:
To evaluate the effect of weight loss on vascular function in obese with poor cardiovascular health. The investigators will evaluate the effects of weight loss on total and central body adiposity, blood pressure, central hemodynamic parameters, arterial stiffness, endothelial function, apnea-hypopnea index, insulin resistance and inflammatory markers.

DETAILED DESCRIPTION:
Excessive adipose tissue is associated with adverse metabolic effects and is an important risk factor for chronic diseases. According to the American Heart Association, most cardiovascular events can be prevented by adhering to healthy practices, reflecting cardiovascular health as poor, intermediate, and ideal. Methods: Both sexes, aged between 40 and 70 years, with body mass index ≥ 30 and < 40 kg/m² will be included and clinical, anthropometric, body composition and laboratory tests will be assessed. In vascular tests, the investigators will evaluate the sympathetic tone using a frequency meter (Polar® RS800), oscillometric pulse wave analysis by Mobil-O-Grah®, post-occlusive microvascular reactivity and carotid ultrasound to measure intimamedia thickness. In the sleep study, the investigators will analyze the presence and degree of obstructive sleep apnea (OSA) through the home polysomnography device (WatchPAT 200®). The first visit will be for screening, clinical and anthropometric evaluation. On the second visit, the vascular tests, instructions and device delivery for sleep study will be performed. Patients will return the following day to return the WatchPAT and to receive the hypocaloric nutritional intervention (800kcal reduction of daily total energy value), which should be followed for 16 weeks. Eight weeks after the beginning of the nutritional intervention a new visit will be scheduled for clinical, nutritional assessment and dietary adjustment. After completing 16 weeks, the patients will return for clinical, laboratory, nutritional, vascular and sleep tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes;
* Age between 40 and 70 years;
* Body mass index (BMI) ≥ 30 kg/m² and <40 kg/m².

Exclusion Criteria:

* Systolic blood pressure ≥ 160 and/or diastolic blood pressure ≥ 100 mmHg;
* Diabetes mellitus; Hormone replacement therapy;
* Evidence of secondary hypertension;
* Clinically evident changes in thyroid function;
* Acute or chronic kidney or liver disease;
* History of cancer in the last 5 years;
* Clinically evident coronary disease with a history of acute myocardial infarction and/or myocardial revascularization, clinical signs of heart failure, cardiac arrhythmia or clinically significant valve disease;
* Previous stroke;

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-21 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2023-11-20 (Estimated)

PRIMARY OUTCOMES:
Pulse wave velocity | Change in PWV after 16-week dietary intervention
  Pulse wave velocity (PWV) will be evaluated by oscillometric monitoring system via Mobil-O -Graph®

SECONDARY OUTCOMES:
Endothelial function | Change in endothelial function after 16-week dietary intervention
  Microvascular reactivity will be evaluated using the laser system contrast image (LSCI)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle R Cunha, MSc, Principal Investigator — Rio de Janeiro State University; Samanta S Mattos, MSc, Principal Investigator — Rio de Janeiro State University
Locations (2):
- Brazil (2):
  - Hospital Universitario Pedro Ernesto, Rio de Janeiro
  - Rio de Janeiro State University, Rio de Janeiro

IPD SHARING:
Plan to Share IPD: No